CLINICAL TRIAL: NCT04332978
Title: Prospective, Comparative, Double-blind, Parallel, Multicentric, Randomized Study Between Two Brands of Fluticasone Propionate Nasal Topic in The Control of Perene Allergic Rhinithis Symptoms
Brief Title: Topical Nasal Fluticasone Propionate in the Control of Allergic Rhinitis SymptomsPerene
Acronym: LB1108
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LB1108
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Plurair; Fluoticasone propionate; topic; nasal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Fluticasone

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, comparative, double-blind, parallel, multicenter, randomized, non-inferiority clinical study between two brands of nasal topical fluticasone propionate:
  * Plurair® - Experimental medicine.
  * Flixonase® - Comparator. Study treatment was allocated by centralized randomization, and each participant remained on the same treatment (dose, dosing regimen and brand) allocated throughout the study period.
Who Masked: Participant, Investigator
Masking Description: In the present double-blind study, the original bottles of the two drugs under study (Plurair® and Flixonase®) had their labels sealed and were packed in identical secondary packaging (with specific label for clinical research), associated with a unique identification code.
  Page 75 of 207 Clinical Report LB1108 Version 1.0 of February 8, 2018 CONFIDENTIAL Libbs Farmacêutica Ltda. Each cartridge of the study drug had a unique identification code related to one of the treatment arms through an electronically generated list, stratified by center. Participants were allocated to one of two treatment groups at a 1: 1 ratio. This list was not accessible to the study doctor, study participant and team, in order to guarantee the study blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Drug names: Fluticasone Propionate - PLURAIR® brand Pharmaceutical form: Nasal spray (50mcg / dose) Administration: Topical nasal route Posology 02 jets in each nostril 1 time a day - Single daily topical nasal dose of 200 mcg / day (2 jets / nostril = 100 mcg / nostril), preferably in the morning, upon waking up and at the same time, for 4 weeks.
  Manufacturer: Libbs Farmacêutica Ltda. Presentation: Deliver 1 bottle of 120 doses in original packaging
  Interventions: Drug: Fluticasone Propionate
- Group II (Active Comparator): Fluticasone Propionate - FLIXONASE® brand Nasal spray (50mcg / dose) Topical nasal route 02 jets in each nostril once a day - Single daily topical nasal dose of 200 mcg / day (2 jets / nostril = 100 mcg / nostril), preferably in the morning, upon waking up and at the same time, for 4 weeks.
  GlaxoSmithKline. Deliver 1 bottle of 120 doses in original packaging
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate

SUMMARY:
Phase III Study to Demonstrate the non inferiority of PLURAIR® branded nasal topical Fluticasone Propionate (FP) in relation to the FLIXONASE® brand reference drug in the control of nasal symptoms related to perennial allergic rhinitis.

DETAILED DESCRIPTION:
This study was conducted to demonstrate the non inferiority of the topical nasal fluticasone propionate of the brand Plurair® in relation to the reference drug Flixonase® in the control of symptoms related to perennial allergic rhinitis. Allergic rhinitis is one of the most common forms of non-infectious rhinitis, characterized mainly by symptoms such as sneezing, runny nose and nasal congestion. Depending on the time of exposure to allergens and the duration of symptoms, allergic rhinitis is classified as perennial (OKUBO, 2009).

Studies for the assessment of perennial allergic rhinitis through symptom analysis used diaries provided to the participants, so that they could describe their symptoms, starting in the screening phase and ending at the end of treatment. In the present study, participants recorded, in the diary, the severity of their rhinitis symptoms (obstruction, runny nose, nasal itching and sneezing) and also associated eye symptoms (watery eyes, itchy eyes and redness) using a four-point scale (0-absent, 1-mild, 2-moderate and 3-severe). For the purpose of analyzing the primary parameter, the total daily reflective nasal symptoms (NRT) was obtained by averaging the total morning and evening scores for each day ([morning NRT + night NRT] / 2) of the individual nasal symptoms - obstruction, itching, runny nose and sneezing - assessed reflexively in the last 12 hours.

This study in its design and analysis of efficacy and safety followed the guidelines of regulatory agencies in the United States of America (FDA, 2000) and Canada (CANADA HEALTH, 2011).

Fluticasone propionate is a potent intranasal corticosteroid with negligible bioavailability, effective in the treatment of nasal symptoms of allergic rhinitis. The onset of the therapeutic effect of fluticasone propionate occurs within 12 hours when 200 μg of the medication is administered once a day (RATNER, 2008).

Following guidelines for the use of fluticasone propionate and guidelines for the assessment of symptoms of perennial allergic rhinitis, the objective of the present clinical study was to evaluate the efficacy and safety of two formulations of fluticasone propionate as a single agent in the treatment of perennial allergic rhinitis through relief of nasal symptoms assessed by recording in the participants' symptom diary.

This study was conducted in accordance with the proposal for the treatment of perennial allergic rhinitis, with local clinical research regulations, with the International Harmonization Conference (ICH) Good Clinical Practices and with the principles of the Declaration Helsinki and their respective revisions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 12 years and <60 years old on the date of the selection visit;
* Clinical history suggestive of perennial allergic rhinitis for at least 02 years;
* Atopy proved through positive evaluation for at least one inhaled allergen (valid positive RAST test performed up to 12 months before the date of the selection visit - or positive Phadiatop® ** performed during the selection period);
* Present the score for reflective nasal symptoms (runny nose, nasal itching, nasal obstruction and sneezing) equal to or greater than the average of 12 points out of a total of 24, during the 4 days preceding the randomization visit OR Present a score of reflective nasal symptoms (runny nose, itchy nose, nasal obstruction and sneezing) at least 12, for at least 4 days, not necessarily consecutive, within a seven-day selection period;
* "Research participant's diary - selection" correctly filled out, considering at least 80% of the completed information regarding nasal and ocular symptoms in the two periods (morning and night);
* Availability of telephone contact for follow-up;
* Signature of the Free and Informed Consent Term and Free and Informed Consent Term, when applicable.

Exclusion Criteria:

* Pregnancy or lactation;
* Women who declare that they have the potential to become pregnant and do not want to adopt any contraceptive method, including: sexual abstinence, mechanical barrier, IUD, oral contraceptive, injectable contraceptive, hormonal implant, hormonal transdermal patch, prior sterilization, etc;
* Other clinical forms of rhinitis: seasonal allergic, medication, vasomotor, atrophic, etc;
* History compatible with IVAS or acute sinusitis in the 15 days prior to the selection visit, symptomatic chronic sinusitis, nasal polyposis;
* Concomitant cardiovascular / hepatic / pulmonary / renal / neurological / neoplastic disease and others, which medical criteria may compromise the patient's participation in the study;
* Current smoking or previous smoking for less than 3 months;
* Cataract, glaucoma, herpes simplex ocular;
* Asthma, with the exception of controlled conditions (GINA Criteria - Global Initiative for Asthma - modified: absence of daytime symptoms, nighttime despair and experiences in experimental activities) without the need for specific medication;
* Previous use of:
* Antihistamine for less than 10 days with the exception of azelastine / astemizole for less than 12 weeks.
* Topical, intranasal and systemic corticosteroids for less than 4 weeks;
* Antileukotriene / anticholinergic / antifungal / antibiotics less than 7 days ago
* Intranasal or systemic decongestant for less than 03 days;
* Non-hormonal anti-inflammatory, including acetylsalicylic acid with use in less than 10 days;
* Use of drugs with the potential to alter cytochrome P450 (eg, ritonavir and ketoconazole, but not exclusively) or with possible clinical influence (eg, tricyclic antidepressants, but not exclusively) or with nasal administration (eg, insulin, but not exclusively);
* History of nasosinusal surgery;
* Results of laboratory selection tests with significant clinical changes (complete blood count, TGO / AST, TGP / ALT, salt, potassium, urea, creatinine, fasting glucose and serum cortisol), which a doctor may compromise the patient's participation in. study;
* Serious illness or condition that the doctor may compromise the patient's participation in the study.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 566 (Actual)
Dates: Start 2014-07-04; Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Variation of the mean of total reflective nasal symptoms (TSNr) | daily records over the 4 weeks of treatment in relation to their baseline value.
  Patients should be instructed to classify and note the severity of nasal symptoms (itching, sneezing, obstruction and coryza) using the "Research participant's diary", the reflexive way in the last 12 hours, with an assessment in the morning and another at night (twice a day, regardless of specified times), with a 4-point scale below:
  0: ABSENT - this symptom is not present.
  1. Mild - this symptom is present, but does not bother.
  2. MODERATE - this symptom is present and is substantially received, but it does not get in the way of your daily activities / sleep quality.
  3. SEVERE - this symptom is present, enters substantially and gets in the way of your daily activities / sleep quality.

SECONDARY OUTCOMES:
Variation of total instant nasal symptoms (TSNi) | over the 4 weeks of treatment
  Patients should be instructed to classify and note the severity of nasal symptoms (itching, sneezing, obstruction and runny nose) individually in the "Research participant's diary", instantly in the morning (upon waking up and before using the medication, without consideration) specific times), according to the 4-point scale below:
  0: ABSENT - this symptom is not present.
  1. Mild - this symptom is present, but does not bother.
  2. MODERATE - this symptom is present and substantially bothers, but it does not get in the way of your daily activities / sleep quality.
  3. SEVERE - this symptom is present, it substantially bothers and gets in the way of your daily activities / sleep quality.
Variation of each nasal symptom | over the 4 weeks of treatment
  Patients should be instructed to classify and note the severity of nasal symptoms (itching, sneezing, obstruction and runny nose) individually in the "Research participant's diary", in a reflexive way in the last 12 hours, with an assessment in the morning and another in the evening (twice a day, regardless of specific times), according to the 4-point scale below:
  0: ABSENT - this symptom is not present.
  1. Mild - this symptom is present, but does not bother.
  2. MODERATE - this symptom is present and substantially bothers, but it does not get in the way of your daily activities / sleep quality.
  3. SEVERE - this symptom is present, it substantially bothers and gets in the way of your daily activities / sleep quality.
Variation of total ocular symptoms and in each specific ocular symptom | over the 4 weeks of treatment
  Patients should be instructed to classify and note the severity of eye symptoms individually - tearing, itching and redness - in the "Research participant's diary", in a reflexive way in the last 12 hours, with an assessment in the morning and another at night (two times a day, without considering specific times), according to the 4-point scale below:
  0: ABSENT - this symptom is not present.
  1. Mild - this symptom is present, but does not bother.
  2. MODERATE - this symptom is present and substantially bothers, but it does not get in the way of your daily activities / sleep quality.
  3. SEVERE - this symptom is present, it substantially bothers and gets in the way of your daily activities / sleep quality.
Patient's overall impression of treatment efficacy at the end of the study | over the 4 weeks of treatment
  At the end of treatment (4 weeks), each patient should assess their overall satisfaction with the treatment's effectiveness, according to the following scale:
  0 = complete improvement of symptoms
  1. = moderate symptom improvement
  2. = slight improvement of symptoms
  3. = no change in symptoms
  4. = slight worsening of symptoms
  5. = moderate worsening of symptoms
  6. = severe worsening of symptoms
Researcher's general impression at the end of the study | over the 4 weeks of treatment
  At the end of the treatment (4 weeks), the researcher will answer about his general impression regarding the effectiveness of the treatment, according to the following scale:
  0 = complete improvement of symptoms
  1. = moderate symptom improvement
  2. = slight improvement of symptoms
  3. = no change in symptoms
  4. = slight worsening of symptoms
  5. = moderate worsening of symptoms
  6. = severe worsening of symptoms